CLINICAL TRIAL: NCT00742326
Title: Pioglitazone for Hepatic Steatosis in HIV/HCV Co-infection
Brief Title: Pioglitazone to Treat Fatty Liver in Patients With HIV and Hepatitis C Infections
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment stopped prior to complete enrollment due to slow accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 080201
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: HIV; Hepatitis C; Liver Disease; Fatty Liver; Steatosis
Keywords: HIV; Hepatitis C; Liver Disease; Fatty Liver; Steatosis
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Fatty Liver | interventions — Pioglitazone; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental): pioglitazone 45 mg daily for 48 weeks
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): one capsule daily for 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — 45 mg/daily
  Other Names: Avandia
  Arms: Pioglitazone
Drug: Placebo — one capsule daily
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of pioglitazone in reducing liver fat content in patients with HIV and hepatitis C virus (HCV) infections. Fatty liver and accompanying insulin resistance in patients with HIV and HCV co-infections is associated with inflammatory changes, liver fibrosis and a poorer response to HCV treatment. Pioglitazone is a drug that helps to reduce the body's resistance to insulin. It is approved by the Food and Drug Administration to treat diabetes.

Patients with HIV and HCV co-infections who have hepatic steatosis (fatty liver) may be eligible for this study. Candidates are screened with a medical history and physical examination, blood and urine tests, magnetic resonance imaging (MRI) of the liver to measure liver fat and, if needed, a liver biopsy to confirm the diagnosis of liver steatosis.

* Participants are randomly assigned to take either pioglitazone therapy or placebo for 48 weeks. This is followed by a second 48-week treatment period in which all participants take pioglitazone.
* There are approximately 12 visits during the 96 weeks of the study. Participants will receive a physical assessment, blood and urine tests at each visit. In addition, periodic assessments of dietary habits, body composition, oral glucose tolerance testing, and health related quality of life questionnaires will be completed.
* A repeat MRI of the liver is performed at 48 weeks and at the end of the study to evaluate any potential changes in liver fat and inflammation. In addition, there is a follow-up liver biopsy at 48 weeks and an optional liver biopsy at 96 weeks.

DETAILED DESCRIPTION:
Following the introduction of effective antiretroviral therapy for HIV, the management of co-morbidities such as hepatitis C virus (HCV) has taken on increasing significance in the care and health maintenance of chronically infected patients. HCV co-infection is common in HIV, with an estimated prevalence of 30 percent among HIV-infected adults in the US. Further, the reported prevalence of hepatic steatosis in HIV/HCV co-infection is between 40-67 percent.

In recent years, the significance of hepatic steatosis and accompanying insulin resistance in HCV has gained increasing recognition. For example, steatosis is associated with increased rates of necro-inflammatory change and fibrosis in HIV/HCV co-infected patients. Furthermore, studies showed that, among non-HIV infected HCV patients, the presence of steatosis and/or insulin resistance was associated with poorer response to HCV therapy. These observations have led to research interest in treating hepatic steatosis in HCV, particularly in the context of pegylated interferon and ribavirin therapy.

Administration of the thiazolidinedione, pioglitazone, leads to significant reductions in hepatic steatosis, inflammation and in some cases fibrosis in patients with non-alcoholic steatohepatitis (NASH). Therefore, the potential benefits of pioglitazone therapy in the setting of HIV/HCV co-infection and hepatic steatosis will be determined. The proposed study is a 48-week, double-blind, randomized placebo-controlled trial of pioglitazone (45 mg/day) in 50 HIV/HCV-infected men and women. After the 48-week randomized portion of the trial, all participants will enter a 48-week open treatment extension arm irrespective of original randomization. It is anticipated that 100 subjects will be needed to be screened to identify a sufficient number of eligible participants to enroll in the study.

The primary outcome variable of interest in this trial will be the change in hepatic fat content measured by magnetic resonance (MR) spectroscopy. Important secondary outcomes will be histologic improvement on liver biopsy performed at baseline and 48 weeks, as well as improvements in transaminase levels and insulin resistance. The open treatment extension will allow all participants an opportunity to receive active study medication and it will allow the potential benefits of additional pioglitazone therapy to be assessed. In this way, important information about the efficacy of pioglitazone to treat hepatic steatosis and improve the metabolic profile in HIV/HCV co-infected patients will be obtained.

ELIGIBILITY:
* INCLUSION CRITERIA:

Men and women, 18 years of age or greater

Confirmed HIV infection by ELISA and Western blot

No changes in antiretroviral regimen within the prior 3 months--Individuals not currently taking antiretroviral therapy will be eligible. Individuals requiring medically indicated adjustments of antiretroviral therapy during the course of the study will be eligible.

Confirmed HCV infection, and no current or recent (within the past 3 months) HCV treatment and no plans to start HCV antiviral therapy in the foreseeable future.

H-MRS liver fat content greater than 5 percent and confirmed steatosis on liver biopsy within 1 year

Fasting glucose less than 126 mg/dL

Platelets greater than or equal to 75,000/uL; INR less than 1.6

Willingness to avoid medications and herbal supplements which may increase the risk of bleeding for one week prior to and one week following liver biopsy (e.g. aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), Vitamin E, fish oil and gingko biloba).

Willingness to restrict physical activity 72 hours after liver biopsy

If premenopausal female, willingness to use 2 forms of effective birth control on this study to avoid pregnancy.

Have a primary care physician

Willingness to have specimens stored.

EXCLUSION CRITERIA:

Current thiazolidinedione use or use in the last 6 months, known allergy or sensitivity to a thiazolidinedione

Use of insulin or other oral hypoglycemics, or known diabetes

Current pregnancy, breast feeding, or pregnancy within the past 6 months or desire to become pregnant within the next 2 years.

Child-Pugh-Turcotte (CPT) score greater than class A

ALT greater than 4 times the upper limit of normal

Current or history of heart failure (New York Heart Association [NYHA] Class III or IV cardiac status)

Hemoglobin level less than 9g/dL

Active or ongoing infection with Hepatitis A or B

Known or suspected liver disease such as autoimmune hepatitis, Wilson's disease, alpha-1-antitrypsin deficiency, cystic fibrosis, hemochromatosis, glycogen storage disease, amyloidosis, primary biliary cirrhosis, sclerosing cholangitis, or any primary or secondary hepatic tumor

Current alcohol/substance abuse

Use of growth hormone, prednisone or other anabolic agents (except for physiologic testosterone replacement) currently or within the past 3 months. One day or less of corticosteroid within the prior 90 days of screening is allowed as is stable dose inhalation corticosteroids

Concurrent use of ketoconazole

Active opportunistic infection (except thrush) or neoplasm (except Kaposi's sarcoma, skin cancer, cancer of the cervix or anus)

Any known contraindications to percutaneous liver biopsy including elevated PT/PTT

Severe psychiatric illness that would interfere with adherence to protocol requirements

Current treatment with interleukin-2, interferon-alpha, or other investigational agent(s) within the past 6 months (This does not pertain to ARVs obtained through expanded access)

Any significant medical condition for which the investigator believes a liver biopsy or participation in the research protocol may be contraindicated

Any contraindication to MRI scan, including excess body size

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen M Hadigan, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - VA Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Decision will be made at the time of request

REFERENCES:
- [Background] Jain MK, Skiest DJ, Cloud JW, Jain CL, Burns D, Berggren RE. Changes in mortality related to human immunodeficiency virus infection: comparative analysis of inpatient deaths in 1995 and in 1999-2000. Clin Infect Dis. 2003 Apr 15;36(8):1030-8. doi: 10.1086/368186. Epub 2003 Apr 2. PMID 12684916
- [Background] Sulkowski MS, Mast EE, Seeff LB, Thomas DL. Hepatitis C virus infection as an opportunistic disease in persons infected with human immunodeficiency virus. Clin Infect Dis. 2000 Apr;30 Suppl 1:S77-84. doi: 10.1086/313842. PMID 10770916
- [Background] Sulkowski MS, Mehta SH, Torbenson M, Afdhal NH, Mirel L, Moore RD, Thomas DL. Hepatic steatosis and antiretroviral drug use among adults coinfected with HIV and hepatitis C virus. AIDS. 2005 Mar 24;19(6):585-92. doi: 10.1097/01.aids.0000163935.99401.25. PMID 15802977
- [Background] Matthews L, Kleiner DE, Chairez C, McManus M, Nettles MJ, Zemanick K, Morse CG, Benator D, Kovacs JA, Hadigan C. Pioglitazone for Hepatic Steatosis in HIV/Hepatitis C Virus Coinfection. AIDS Res Hum Retroviruses. 2015 Oct;31(10):961-6. doi: 10.1089/AID.2015.0093. Epub 2015 Aug 24. PMID 26214341

RESULTS

PARTICIPANT FLOW:
Groups:
- Pioglitazone: pioglitazone 45 mg daily for 48 weeks
  Pioglitazone
- Placebo: Placebo once daily for 48 weeks
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (5) | 53 (6) | 52 (6)
Gender [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 6 | 12
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Steatosis and Hepatic Inflammation/Fibrosis in HIV/HCV Co-infected Patients With Steatosis.
Description: Change in hepatic steatosis and hepatic inflammation/fibrosis in HIV/HCV co-infected patients with steatosis. Change in Hepatic Fat Content measured by MR spectroscopy: 48 weeks compared to Baseline
Time Frame: 48 weeks
Population: Two subjects (one in each group) did not have a follow up MRI for comparision to baseline. One developed claustrophobia and could not tolerate MRI and one was discontinued from study due to other illnesses.
Measure: Mean (Standard Deviation); unit: percentage of hepatic fat on MRS
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 5 | 6
percentage of hepatic fat on MRS | -7.43 (4.6) | -2.17 (9.9)

2. Secondary Outcome: Change in Insulin Resistance in HIV- and HCV-infected Patients With Steatosis Compared to Placebo
Description: Change in Glucose Area Under the Curve from standard oral glucose challenge ( baseline to 2 hours): Week 48 - Baseline values
Time Frame: 48 weeks
Population: One subject in the placebo arm was discontinued due to health issues and does not have a 48 week OGTT available
Measure: Mean (Standard Deviation); unit: mg*120 minutes/dL
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 6 | 6
mg*120 minutes/dL | -31 (29.2) | 11 (43.5)

ADVERSE EVENTS:
Time Frame: 48 weeks of randomized study participation
Arm/Group | Pioglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/7
Other Adverse Events (participants affected / at risk) | 3/6 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=6) | Placebo (N=7)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Patient was diagnosed with advanced stage lung cancer during study participation. Participation in the study was discontinued by the study team when the diagnosis was made.
Dental Abscess (Infections and infestations) | 0 (0) | 1 (1) — Dental abscess requiring treatment related to poor dentition
Renal Insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) — Renal insufficiency identified, related to HIV antiretroviral therapy. Resolved after changing antiretroviral mediactions
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=6) | Placebo (N=7)
Fatigue (General disorders) | 1 (6) | 2 (7)
Weight Gain (Metabolism and nutrition disorders) | 2 (6) | 1 (7)
Decrease serum albumin (Metabolism and nutrition disorders) | 2 (6) | 3 (7)
Increased cholesterol (Endocrine disorders) | 1 (6) | 2 (7)

LIMITATIONS AND CAVEATS:
The study failed to enroll to the originally established sample size due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less